CLINICAL TRIAL: NCT03318354
Title: An Open Label, Randomized, 2-Period, 2-Treatment,2-Sequence, Crossover, Single-Dose BE of Olmesartan Medoxomil Tablets 40 mg [Torrent,India] Versus Benicar 40 mg Tablets [Daiichi Sankyo Inc., USA] in Healthy Subjects-Fasted Condition
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd.'s Olmesartan Medoxomil Tablet Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OLME/10/026
Record Dates: First submitted 2017-10-19; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Torrent's Olmesartan Medoxomil Tablets 40 mg
  Interventions: Drug: Torrent's Olmesartan Medoxomil Tablets 40 mg
- Reference (Active Comparator): Daiichi Sankyo Inc's Benicar Tablets 40 mg
  Interventions: Drug: Daiichi Sankyo Inc's Benicar Tablets 40 mg

INTERVENTIONS:
Drug: Torrent's Olmesartan Medoxomil Tablets 40 mg
  Arms: Test
Drug: Daiichi Sankyo Inc's Benicar Tablets 40 mg
  Arms: Reference

SUMMARY:
Subjects to compare the single dose bioavailability of Torrent's Olmesartan Medoxomil Tablets 40 mg and Benicar 40 mg Tablets of Daichi Sankyo Inc. USA. Dosing periods of studies were separated by a washout period of 7 days.

DETAILED DESCRIPTION:
An Open Label, Randomized, 2-period, 2- Treatment, 2-Sequence, Crossover, Single-dose Bioequivalence Study of Olmesartan Medoxomil Tablets containing Olmesartan Medoxomil 40 mg (Test Formulation, Torrent Pharmaceutical Ltd., India) Versus Benicar® 40 mg Tablets containing Olmesartan Medoxomil 40 mg (Reference, Daiichi Sankyo Inc.,USA) in Healthy Human Volunteers Under Fasting Condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males with age between 18-45 years (both inclusive)
* Weight equal to or more than 50.00 Kgs
* BMI 18.50 - 24.90 Kg/m2
* Healthy as determined by medical history, clinical and laboratory examination performed within 21 days prior to admission day for the first period of the study.
* Must have provided written informed consent for participation in the study in the subject's vernacular language
* In the opinion of the Principal Investigator/Designee, be able to comply with the study procedures and protocol restrictions.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Olmesartan, its excipients or similar classes of drugs
* Any evidence of significant abnormalities upon physical or clinical examination
* Sitting blood pressure less than 100/70 mm Hg or more than 140/90 mm Hg and radical pulse rate less than 60 mm Hg or more than 100 mm Hg per minute at the time of screening.
* Laboratory values, which are significantly different from predefined reference ranges and judged clinically significant.
* Any clinically significant abnormality in ECG.
* Any clinically significant abnormality in Chest X-ray (PA view)
* Regular use of tobacco or nicotine in significant amount in any form (e.g. use of more than 10 cigarettes a day) or have difficulty in abstaining from [smoking] nicotine use for the duration of the study period.
* History of drug dependence or excessive alcohol intake [subjects who drink more than 2 units per day (30 ml of 40% alcohol) or more than 14 units per week] on a habitual basis, or inability to abstain from alcohol for the duration of study period.
* History or presence of serious gastrointestinal, liver, kidney, heart, lung, neurological or blood disease, diabetes or glaucoma.
* History or presence of any chronic illnesses such as arthritis, asthma, epilepsy, hypertension etc.
* Presence of disease markers of HIV 1 OR 2, Hepatitis B or C Viruses and VDRL.
* Positive result for drug(s) of abuse testing (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opioids) in urine.
* Positive test for alcohol breath analyzer test.
* History and presence of any psychiatric illness.
* History and presence of any illness including allergic skin diseases, allergic asthma and drug-induced allergy, e.g. NSAIDs
* History of significant blood loss (≥ 350 mL) due to any reason, including blood donation within last 12 weeks prior to screening.
* Existence of any surgical or medical condition which in the judgment of Principal Investigator/ Designee might interfere with the absorption, distribution, metabolism or excretion of the study drug, or, is likely to compromise the safety of subject.
* Intake of any enzyme-modifying drugs such as cimetidine, theophylline, benzodiazepines, ranitidine, proton pump inhibitors, erythromycin, diuretics, ketoconazole, anti hypertensive drugs, dopamine agonists, etc within 30 days of study drug administration, or administration/ intake of any prescription or OTC drug including vitamins and natural supplements within 30 days of study drug administration. In such cases, enrolment of the subject in the study will be at the discretion of the Principal Investigator/designee.
* Intake of unusual diet (e.g. low sodium) for two weeks prior to screening and throughout the subject's participation the study. In such case, subject selection will be at the discretion of the Principal investigator/ designee.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre dose to 72 hours post dose.
AUC | Pre dose to 72 hours post dose.

IPD SHARING:
Plan to Share IPD: No